CLINICAL TRIAL: NCT05874674
Title: The Safety of Nafamostat Mesylate for Patients With High Risk Bleeding Diathesis Undergoing Hemodialysis: A Pilot Study
Brief Title: The Safety of Nafamostat Mesylate for Patients With High Risk Bleeding Undergoing Hemodialysis: A Pilot Study
Acronym: Nafamostat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CR122018
Record Dates: First submitted 2023-04-18; First posted 2023-05-25 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Dialysis; Complications; Bleeding
Keywords: dialysis; bleeding; nafamostat; heaprin
MeSH Terms: conditions — Hemorrhage | interventions — nafamostat

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nafamostat (Active Comparator): Patients received dialysis through nafamostat
  Interventions: Drug: Nafamostat Mesylate
- Cnoxane (No Intervention): Patients received dialysis through cnoxan

INTERVENTIONS:
Drug: Nafamostat Mesylate — Comparison effect of nafamostat and cnoxan
  Other Names: cnoxan
  Arms: nafamostat

SUMMARY:
Comparison nafamostat and low molecular weight heparin among dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* platelet below 10k PTT above 60 second INR above 20 patient with bleeding (epistaxis, orbital bleeding, hematuria) recent brain hemorrhage (within 6 months) receiving anticoagulant therapy (coumadin or NOAC) dual antiplatelet agent users received major surgery within one month

Exclusion Criteria:

* cancer liver cirrhosis pregnancy drug allergy current bleeding on major organ (brain, gastrointestinal)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with severe bleeding | 6 month
  Brain hemorrhage (on brain CT), gastrointestinal bleeding (on EGD)

SECONDARY OUTCOMES:
Number of patients with dialysis circuit clot | 6 month
  Dialysis circuit clotting due to not enough anticoagulation

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Unviersity Wonju College of Medicin, Wŏnju, Kangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593